CLINICAL TRIAL: NCT00013754
Title: Child Environmental Health Center--Reducing Pesticide Exposure in Children of Farmworkers (UW IRB 96-6567-C02, FENSKE, 6/15/00-6/14/01)
Brief Title: Pesticide Exposure Pathways for Farmworker Children
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Collaborators: Environmental Protection Agency (EPA) (U.S. Federal Agency)
Other Study IDs: 9601-CP-001
Record Dates: First submitted 2001-03-29; First posted 2001-03-30 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Poisoning
Keywords: pesticide; insecticide; organophosphate; exposure; child health
MeSH Terms: conditions — Poisoning

SUMMARY:
This project is aimed at better understanding how children living in agricultural environments are exposed to pesticides, and how such exposures can be prevented or reduced. The current project will characterize pesticide exposure pathways for children of farmworkers.

DETAILED DESCRIPTION:
This project is aimed at better understanding how children living in agricultural environments are exposed to pesticides, and how such exposures can be prevented or reduced. Since 1991 our group has investigated pesticide expsoures among children of agricultural families in Washington state, focusing on exposure to organophosphate insecticides. We have demonstrated in these studies that the residential environments of agricultural families have higher pesticide residues than do other homes in this region. We have also found that children living in these residential environments have elevated levels of pesticide metabolites in their urine. We need to better understand how these children are being exposed in order to develop recomendations for exposure prevention or reduction. The current project will characterize pesticide exposure pathways for children of farmworkers. A complementary project is also underway by the UW-Child Health Center to develop and implement a community-wide intervention to reduce the transfer of pesticides from the workplace to the home (take home pathway).

ELIGIBILITY:
Each family recruited must include one child between the ages of 1-5.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2001-03; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Environmental Health, University of Washington, Seattle, Washington, United States